CLINICAL TRIAL: NCT01003639
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study of Weight-Reduction and/or Low Sodium Diet Plus Acetazolamide vs Diet Plus Placebo in Subjects With Idiopathic Intracranial Hypertension With Mild Visual Loss
Brief Title: Idiopathic Intracranial Hypertension Treatment Trial
Acronym: IIHTT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: National Eye Institute (NEI) (NIH); University of Rochester (Other); University of Iowa (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NORDIC01; 1U10EY017281-01A1 (NIH); 1U10EY017387-01A1 (NIH)
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: papilledema; vision loss; headache; obesity; women; diplopia; tinnitus
MeSH Terms: conditions — Pseudotumor Cerebri; Papilledema; Vision Disorders; Headache; Obesity; Diplopia; Tinnitus | interventions — Acetazolamide; Naproxen; Acetaminophen; Aspirin; Ibuprofen; Codeine; butalbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide given in escalating doses
  Interventions: Drug: Acetazolamide; Behavioral: Formal weight loss counselling program
- Sugar pill (Placebo Comparator): Given in escalating "dose" (number of pill)
  Interventions: Drug: Placebo; Behavioral: Formal weight loss counselling program

INTERVENTIONS:
Drug: Acetazolamide — Subjects will begin with four 250 mg tablets daily. Tablets will be divided among two doses, taken with meals. Beginning on day 7, subjects will increase the dose by 1 pill every week until 16 tablets daily is reached (4 grams acetazolamide or placebo) or side effects prohibit increasing the dosage further. Thus, subjects who are able to tolerate the study medication will reach the maximum dose by day 84.
  Other Names: naproxen; acetaminophen; aspirin; ibuprofen; codein; butalbital
  Arms: Acetazolamide
Drug: Placebo — Subjects will begin with four tablets daily. Tablets will be divided among two doses, taken with meals. Beginning on day 7, subjects will increase the dose by 1 pill every week until 16 tablets daily is reached (4 grams acetazolamide or placebo) or side effects prohibit increasing the dosage further. Thus, subjects who are able to tolerate the study medication will reach the maximum dose by day 84.
  Other Names: naproxen; acetaminophen; aspirin; ibuprofen; codein; butalbital
  Arms: Sugar pill
Behavioral: Formal weight loss counselling program — Teleconference, web-based from central location, using site visits and subject self-assessment tools
  Other Names: naproxen; acetaminophen; aspirin; ibuprofen; codein; butalbital

SUMMARY:
Idiopathic intracranial hypertension (IIH), also called pseudotumor cerebri, is a disorder of elevated intracranial pressure of unknown cause [Corbett, et al., 1982; Wall, et al., 1991]. Its incidence is 22.5 new cases each year per 100,000 overweight women of childbearing age, and is rising [Garrett, et al., 2004] in parallel with the obesity epidemic. It affects about 100,000 Americans. Most patients suffer debilitating headaches. Because of pressure on the optic nerve (papilledema), 86% have some degree of permanent visual loss and 10% develop severe visual loss [Wall, et al., 1991]. Interventions to prevent loss of sight, all with unproven efficacy, include diet, diuretics such as acetazolamide, repeated spinal taps, optic nerve sheath fenestration surgery, and cerebrospinal fluid (CSF) shunting procedures. The purported goal of these therapies is to lower intracranial pressure; however, it is unclear which treatments work and by what mechanism. None of these strategies has been verified by properly designed clinical trials. Thus, there is confusion, uncertainty, and weak scientific rationales to guide treatment decisions. This trial will study subjects who have mild visual loss from IIH to (1) establish convincing, evidence-based treatment strategies for IIH to restore and protect vision, (2) follow subjects up to 4 years to observe the long-term treatment outcomes and (3) determine the cause of IIH. To meet those aims, the trial will be divided into a 12-month intervention phase and a 3-year observational phase. Subjects are not required to complete the observational phase of the study, but will be asked to do so and consented for the observational phase of the study at the conclusion of the intervention phase (12 months).

DETAILED DESCRIPTION:
Clinical Phase: Phase II Investigators: NORDIC Network sites Study Centers: 38 study centers Coordinating Center - University of Rochester Statistical Center - University of Rochester Study Period Planned enrollment duration: 2 years Planned duration of treatment: 6 months followed by open-label treatment Planned duration of follow-up: 4.5 years Study Objectives: The primary objective is determining the efficacy of diet plus acetazolamide vs diet alone in reducing or reversing visual loss in subjects with mild visual loss.

The secondary objective is to identify proteomic and genetic risk factors for IIH by screening a large cohort of IIH patients and controls.

Study Population This project will enroll 166 individuals with IIH who are 18-60 years of age. We anticipate that the population will be primarily composed of women in the childbearing years that are overweight. 154 control subjects will also be enrolled. Control subjects will be matched as closely as possibly by age, sex, race, ethnicity and weight to subjects enrolled at the site.

Study Design: Multi-center, double-blind randomized intervention study followed by a 4-year observation period. Subjects will be randomized to diet and acetazolamide or diet and placebo. The study will use 250 mg acetazolamide or matching placebo tablets taken with food at meals and at bedtime. The subject will begin with one tablet four times daily, at meals and at bedtime for the first week. Beginning on Day 7, subjects will increase the dosage by 1 tablet every 4 days until a final dosage of 4 tablets four times daily (4 grams) is reached or side effects prohibit increasing the dosage further. If the study drug is not tolerated at a dose of 250 mg, then 125 mg (1/2 tablet) will be tried. If this is not tolerated, no pharmacologic treatment will be given.

After the 6 month visit, all subjects will transition from study medication to acetazolamide (open label) by replacing one tablet of study drug with 250 mg of acetazolamide every four days. The acetazolamide dose will be titrated in a manner similar to the initial study drug schedule to the maximum tolerated dose of acetazolamide. To avoid treating subjects (who may have initially been assigned to placebo) unnecessarily, any subject with grade 0-1 papilledema will be tapered off study drug but not placed on acetazolamide unless they have persisting headaches or pulse-synchronous tinnitus. If so, they will be placed on acetazolamide regardless of the low papilledema grade. At the 9-month follow-up visit, we will make sure that the subjects' vision is stable after the transition off of study medication. After the 9 month visit, medication will be prescribed by the subject's treating physician. The intervention phase of the study will end at the subject's 12 month visit and subjects will be invited to participate in the observational phase of the study and consented to do so if willing.

Number of Subjects: 166 subjects with IIH and 154 control subjects Main Inclusion Criteria

1. Diagnosis of IIH by modified Dandy criteria
2. Diagnosis of IIH for 6 weeks or less
3. Age 18 to 60 years at time of diagnosis
4. Reproducible visual loss present on automated perimetry (in eye with greatest loss)*
5. perimetric mean deviation (PMD) -2 decibel (dB) up to -5 dB in the worst eye
6. Presence of bilateral papilledema
7. Able to provide informed consent or parental permission with appropriate assent

Main Exclusion Criteria

1. Total treatment of IIH of more than one week in the past six weeks
2. Corticosteroids or surgery used for IIH treatment within the past two months
3. Abnormalities on neurologic examination aside from papilledema and its related visual loss or VI nerve paresis (unless pre-existing and unrelated to IIH)
4. Abnormal CT or MRI scan (intracranial mass, hydrocephalus, dural sinus thrombus or arteriovenous malformation) other than empty sella, dilated optic nerve sheath, flattened sclera, or secondary Chiari
5. CSF pressure less than 200 mm water (patients may have repeat CSF pressure measurements if the first is normal or no opening pressure obtained)
6. Abnormal CSF contents (increased cells, elevated protein, low glucose)
7. Intraocular pressure currently > 28 mm Hg or > 30 mm Hg at any time in the past
8. Refractive error > +/- 6.00 sphere or > +/- 3.00 cylinder in either eye
9. Other disorders causing visual loss except for refractive error and amblyopia including cells in the vitreous or iritis
10. Inability to provide reliable and reproducible visual field examination (failure to maintain fixation using an eye monitoring device, more than 15% false positive errors
11. Abnormal blood work-up indicating a medical or systemic condition associated with raised intracranial pressure (ICP)
12. Exposure to a drug, substance or disorder that has been associated with elevation of intracranial pressure within 2 months of diagnosis such as lithium, vitamin A, tetracycline, steroid withdrawal (see table in Manual of Procedures (MOP) for conditions and drugs)
13. Other condition requiring diuretics, steroids or other pressure lowering agents including topiramate
14. Presence of a medical condition such as renal stones that would contraindicate use of the study drugs (acetazolamide)
15. Pregnancy or unwillingness for subject with childbearing potential to use contraception during the first year of the study
16. Presence of a physical, mental, or social condition likely to affect follow-up (drug addiction, terminal illness, no telephone, homeless)
17. Anticipation of a move from the site area within six months and unwillingness to return for follow-up.

Route and Dosage Form: 250 mg acetazolamide tablets or matching placebo taken with food 4 times daily. Subjects will titrate to a maximum dose of 4 tablets 4 times daily (4 grams) as tolerated. If a subject is not able to tolerate a dose of 250 mg, 125 mg (1/2 tablet) may be tried. If this is not tolerated, no pharmacologic treatment will be given.

Duration of Treatment: 6 months of randomized treatment followed by open label acetazolamide treatment. After the 9-month visit medication will be prescribed by the subject's treating physician. The intervention phase of the study will end at Month 12 and the subject invited to continue in the observational phase.

Primary Outcome Measure(s): The primary outcome measure is the change from baseline to Month 6 in PMD (perimetric mean deviation) in the eye with the most severe initial visual loss.

Secondary Outcome Measure: CSF pressure measurement by lumbar puncture Number of abnormal perimetry test locations Visual field examination ratings (improved, remained the same, or worsened) Papilledema grade QOL assessments Dietary Outcomes (BMI, Waist circumference, urinary sodium) Safety Outcomes: Adverse events will be tabulated by treatment group, severity, and perceived relationship to the study intervention Sample Size Considerations

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IIH by modified Dandy criteria Signs and symptoms of increased intracranial pressure Absence of localizing findings on neurologic examination Absence of deformity, displacement, or obstruction of the ventricular system and otherwise normal neurodiagnostic studies, except for evidence of increased cerebrospinal fluid pressure (>200 mm water). Abnormal neuroimaging except for empty sella turcica, optic nerve sheath enlargement, and smooth-walled non flow-related venous sinus stenosis or collapse106 should lead to another diagnosis Awake and alert No other cause of increased intracranial pressure present
2. Diagnosis of IIH for 6 weeks or less
3. Age 18 to 60 years at time of diagnosis
4. Reproducible visual loss present on automated perimetry (in eye with greatest loss)
5. Average PMD -2 dB up to -5 dB in the worst eye
6. Presence of bilateral papilledema
7. Able to provide informed consent
8. Women of child-bearing potential must use an acceptable form of birth control during the intervention phase of the study. Acceptable forms include oral contraceptives, transdermal contraceptives,

Exclusion Criteria:

1. Total treatment of IIH of more than two weeks (except for acetazolamide which is limited to 1 week). For every day on treatment there must be a one-day washout period.
2. Previous surgery for IIH including optic nerve sheath fenestration, CSF shunting procedures, subtemporal decompression and venous stenting
3. Previous gastric bypass surgery
4. Abnormalities on neurologic examination aside from papilledema and its related visual loss or VI nerve paresis
5. Abnormal CT or MRI scan (intracranial mass, hydrocephalus, dural sinus thrombus or arteriovenous malformation) other than empty sella, unfolded optic nerve sheaths, flattened sclera, or smooth- walled venous stenosis
6. CSF pressure less than 200 mm water (patients may have repeat CSF pressure measurements if the first is normal or no opening pressure obtained)
7. Abnormal CSF contents: increased cells: > 5 cells, elevated protein:

> 45 mg%, low glucose: < 30 mg% (If the lumbar puncture produces a cell count compatible with a traumatic needle insertion, the patient does not need to be excluded if the CSF WBC after correction is 5 wbc/mm3 or less- see Operations Manual for calculation) 8. Intraocular pressure currently > 28 mm Hg or > 30 mm Hg at any time in the past 9. Refractive error > +/- 6.00 sphere or > +/- 3.00 cylinder in either eye with the following exceptions: Subjects with myopia of >-6.00 D sphere but less than or equal to - 8.00 D sphere are eligible if 1)there are no abnormalities on ophthalmoscopy or fundus photos related to myopia that are associated with visual loss (such as staphyloma, retinal thinning in the posterior pole or more than mild optic disc tilt), and 2) the subject wears a contact lens for all perimetry examinations with the appropriate correction. If either the Site Investigator or the PRC director (or his designate) decides there are optic fundus abnormalities of myopia that are associated with visual loss, then 9. Subjects with hyperopia of > +6.00 D but less than or equal to

* 8.00 D sphere are eligible if 1) there is an unambiguous characteristic halo of peripapillary edema as opposed to features of a small crowded disc or other hyperopic change related to visual loss determined by the site investigator or the PRC director (or his designate) and 2) the subject wears a contact le 10. Other disorders causing visual loss except for refractive error and amblyopia including cells in the vitreous or iritis 11. Optic disc drusen on exam or in previous history 12. Presence of diagnosed untreated obstructive sleep apnea 13. Inability to provide reliable and reproducible visual field examination (failure to maintain fixation using an eye monitoring device, more than 15% false positive errors) 14. Abnormal blood work-up indicating a medical or systemic condition associated with raised ICP 15. Study blood results showing severe anemia, leukopenia or thrombocytopenia, renal failure, or hepatic disease, based on the Site Investigator's judgment 16. Type I diabetes or the presence of diabetic retinopathy 17. Exposure to a drug, substance or disorder that has been associated with elevation of intracranial pressure within 2 months of diagnosis such as lithium, vitamin A, various cyclines (see table in Operations Manual for conditions and drugs) 18. Other condition requiring diuretics, oral, I.V. or injectable steroids or other pressure lowering agents including topiramate (nasal, inhaled, or topical steroids are allowed since the systemic effects are small) 19. Presence of a medical condition such as renal stones that would contraindicate use of the study drug (acetazolamide) 20. Pregnancy or unwillingness for subject of childbearing potential to use contraception during the first year of the study 21. Breastfeeding mothers are excluded from participation unless willing to discontinue breastfeeding by the baseline visit 22. Presence of a physical, mental, or social condition likely to affect follow-up (drug addiction, terminal illness, no telephone, homeless) 23. Anticipation of a move from the site area within six months and unwillingness to return for follow-up at an IIHTT study site 24. Allergy to pupil dilating drops or narrow angles precluding safe dilation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wall, MD, Study Director — University of Iowa
Locations (41):
- United States (39):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Doheny Eye Center, University of Southern California, Los Angeles, California
  - The Eye Care Group, PC, Waterbury, Connecticut
  - Bascom Palmer Eye Institute, University of Miami, Miami, Florida
  - Neuro-Ophthamology & Balance Disorders Clinic, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois, Peoria, Illinois
  - Department of Ophthamology and Visual Sciences, University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Greater Baltimore Medical Center Department Of Ophthamology, Baltimore, Maryland
  - Johns Hopkins Universtiy - Wilmer Ophthamological Institute, Baltimore, Maryland
  - Bethesda Neurology, LLC, Bethesda, Maryland
  - Massachusetts Eye and Ear Infirmary - Neuro-Ophthamology Service, Boston, Massachusetts
  - Michigan State University Department of Neurology, East Lansing, Michigan
  - William Beaumont Hosptial Research Institute, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University Eye Institute, St Louis, Missouri
  - University of St. Louis, St Louis, Missouri
  - New Jersey Medical School/University Physicians Associates of New Jersey, Newark, New Jersey
  - New York Eye and Ear Infirmary, New York, New York
  - Weill Cornell Medical College, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - University of Rochester - Flaum Eye Institute, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - SUNY Upstate Medical University, Neurology Medical Service Group, Syracuse, New York
  - Duke Eye Center, Durham, North Carolina
  - Raleigh Neurology Associates, PA, Raleigh, North Carolina
  - Wake Forrest University Eye Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Oregon Health & Science University - Casey Eye Institute, Portland, Oregon
  - University of Pennsylvania, Department of Ophthamology, Philadelphia, Pennsylvania
  - The Methodist Hospital: Methodist Eye Associates, Houston, Texas
  - Universtiy of Houston - University Eye Institute, Houston, Texas
  - University of Texas Science Center, San Antonio, Texas
  - University of Utah, John A. Moran Eye Center, Salt Lake City, Utah
  - University of Virginia - Department of Ophthalmology, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
- Canada (2):
  - University of Calgary: Rockyview General Hospital, Calgary, Alberta
  - Queen's University - Hotel Dieu Hospital, Kingston, Ontario

REFERENCES:
- [Result] NORDIC Idiopathic Intracranial Hypertension Study Group Writing Committee; Wall M, McDermott MP, Kieburtz KD, Corbett JJ, Feldon SE, Friedman DI, Katz DM, Keltner JL, Schron EB, Kupersmith MJ. Effect of acetazolamide on visual function in patients with idiopathic intracranial hypertension and mild visual loss: the idiopathic intracranial hypertension treatment trial. JAMA. 2014 Apr 23-30;311(16):1641-51. doi: 10.1001/jama.2014.3312. PMID 24756514
- [Derived] Wang JK, Kardon RH, Ledolter J, Sibony PA, Kupersmith MJ, Garvin MK; OCT Sub-Study Committee and the NORDIC Idiopathic Intracranial Hypertension Study Group. Peripapillary Retinal Pigment Epithelium Layer Shape Changes From Acetazolamide Treatment in the Idiopathic Intracranial Hypertension Treatment Trial. Invest Ophthalmol Vis Sci. 2017 May 1;58(5):2554-2565. doi: 10.1167/iovs.16-21089. PMID 28492874
- [Derived] Wall M, Thurtell MJ; NORDIC Idiopathic Intracranial Hypertension Study Group. Optic disc haemorrhages at baseline as a risk factor for poor outcome in the Idiopathic Intracranial Hypertension Treatment Trial. Br J Ophthalmol. 2017 Sep;101(9):1256-1260. doi: 10.1136/bjophthalmol-2016-309852. Epub 2017 Jan 27. PMID 28130349
- [Derived] Bruce BB, Digre KB, McDermott MP, Schron EB, Wall M; NORDIC Idiopathic Intracranial Hypertension Study Group. Quality of life at 6 months in the Idiopathic Intracranial Hypertension Treatment Trial. Neurology. 2016 Nov 1;87(18):1871-1877. doi: 10.1212/WNL.0000000000003280. Epub 2016 Sep 30. PMID 27694262
- [Derived] Wall M, Johnson CA, Cello KE, Zamba KD, McDermott MP, Keltner JL; NORDIC Idiopathic Intracranial Hypertension Study Group. Visual Field Outcomes for the Idiopathic Intracranial Hypertension Treatment Trial (IIHTT). Invest Ophthalmol Vis Sci. 2016 Mar;57(3):805-12. doi: 10.1167/iovs.15-18626. PMID 26934136
- [Derived] Sibony PA, Kupersmith MJ; OCT Substudy Group of the NORDIC Idiopathic Intracranial Hypertension Treatment Trial. "Paton's Folds" Revisited: Peripapillary Wrinkles, Folds, and Creases in Papilledema. Ophthalmology. 2016 Jun;123(6):1397-9. doi: 10.1016/j.ophtha.2015.12.017. Epub 2016 Jan 14. No abstract available. PMID 26778344
- [Derived] Cello KE, Keltner JL, Johnson CA, Wall M; NORDIC Idiopathic Intracranial Hypertension Study Group. Factors Affecting Visual Field Outcomes in the Idiopathic Intracranial Hypertension Treatment Trial. J Neuroophthalmol. 2016 Mar;36(1):6-12. doi: 10.1097/WNO.0000000000000327. PMID 26618282
- [Derived] Sibony PA, Kupersmith MJ, Feldon SE, Wang JK, Garvin M; OCT Substudy Group for the NORDIC Idiopathic Intracranial Hypertension Treatment Trial. Retinal and Choroidal Folds in Papilledema. Invest Ophthalmol Vis Sci. 2015 Sep;56(10):5670-80. doi: 10.1167/iovs.15-17459. PMID 26335066
- [Derived] Fischer WS, Wall M, McDermott MP, Kupersmith MJ, Feldon SE; NORDIC Idiopathic Intracranial Hypertension Study Group. Photographic Reading Center of the Idiopathic Intracranial Hypertension Treatment Trial (IIHTT): Methods and Baseline Results. Invest Ophthalmol Vis Sci. 2015 May;56(5):3292-303. doi: 10.1167/iovs.15-16465. PMID 26024112
- [Derived] OCT Sub-Study Committee for NORDIC Idiopathic Intracranial Hypertension Study Group; Auinger P, Durbin M, Feldon S, Garvin M, Kardon R, Keltner J, Kupersmith MJ, Sibony P, Plumb K, Wang JK, Werner JS. Baseline OCT measurements in the idiopathic intracranial hypertension treatment trial, part II: correlations and relationship to clinical features. Invest Ophthalmol Vis Sci. 2014 Nov 4;55(12):8173-9. doi: 10.1167/iovs.14-14961. PMID 25370513
- [Derived] OCT Sub-Study Committee for NORDIC Idiopathic Intracranial Hypertension Study Group; Auinger P, Durbin M, Feldon S, Garvin M, Kardon R, Keltner J, Kupersmith M, Sibony P, Plumb K, Wang JK, Werner JS. Baseline OCT measurements in the idiopathic intracranial hypertension treatment trial, part I: quality control, comparisons, and variability. Invest Ophthalmol Vis Sci. 2014 Nov 4;55(12):8180-8. doi: 10.1167/iovs.14-14960. PMID 25370510
- [Derived] Keltner JL, Johnson CA, Cello KE, Wall M; NORDIC Idiopathic Intracranial Hypertension Study Group. Baseline visual field findings in the Idiopathic Intracranial Hypertension Treatment Trial (IIHTT). Invest Ophthalmol Vis Sci. 2014 Apr 29;55(5):3200-7. doi: 10.1167/iovs.14-14243. PMID 24781936
- [Derived] Wall M, Kupersmith MJ, Kieburtz KD, Corbett JJ, Feldon SE, Friedman DI, Katz DM, Keltner JL, Schron EB, McDermott MP; NORDIC Idiopathic Intracranial Hypertension Study Group. The idiopathic intracranial hypertension treatment trial: clinical profile at baseline. JAMA Neurol. 2014 Jun;71(6):693-701. doi: 10.1001/jamaneurol.2014.133. PMID 24756302
- See also: Organization Web-site — http://NORDICclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 38 academic and private practice sites in North America from March 2010 to November 2012,with follow-up ending in June 2013.
Pre-assignment Details: Randomization was stratified by site and included blocking to ensure balance among the treatment groups within a site after every 4 participants had been enrolled at that site.
Groups:
- Acetazolamide: Acetazolamide given in escalating doses
  Acetazolamide: Subjects will begin with four 250 mg tablets daily.
- Sugar Pill: Given in escalating "dose" (number of pill)
  Placebo: Subjects will begin with four tablets daily.
Period: Overall Study
Arm/Group | Acetazolamide | Sugar Pill
Started | 86 | 79
Completed | 69 | 57
Not Completed | 17 | 22
Not completed — Lost to Follow-up | 6 | 9
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Lack of Efficacy | 1 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide | Sugar Pill | Total
Number analyzed (Participants) | 86 | 79 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.9) | 30.0 (8.0) | 29.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 77 | 161
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 16 | 41
  White | 54 | 54 | 108
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 3 | 7 | 10
Weight [Mean (Standard Deviation); unit: kg] | 108.1 (25.6) | 107.3 (24.5) | 107.7 (25.0)
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] — Body mass index is calculated as weight in kilograms divided by height in meters squared.
  Kg/m^2 | 40.0 (8.5) | 39.9 (8.1) | 39.9 (8.3)
Weight change in the past 6 mo [Mean (Standard Deviation); unit: kg] | 10.7 (16.7) | 8.8 (16.9) | 9.8 (16.7)
Transient visual obscurations [Number; unit: participants]
  yes | 55 | 57 | 112
  No | 31 | 22 | 53
Diplopia [Number; unit: participants]
  Yes | 20 | 16 | 36
  No | 66 | 63 | 129
Constant visual loss [Number; unit: participants]
  Yes | 25 | 28 | 53
  No | 61 | 51 | 112
Photophobia [Number; unit: participants]
  Yes | 42 | 37 | 79
  No | 44 | 42 | 86
Headache [Number; unit: participants]
  Yes | 70 | 69 | 139
  No | 16 | 10 | 26
Pulsatile tinnitus [Number; unit: participants]
  Yes | 45 | 41 | 86
  No | 41 | 38 | 79
Perimetric mean deviation [Mean (Standard Deviation); unit: dB] — Perimetric mean deviation is a measure of global visual field loss (mean deviation from age-corrected normal values), with a range of 2 to -32 dB; larger negative values indicate greater vision loss.
  dB
    Study eye | -3.5 (1.2) | -3.5 (1.1) | -3.5 (1.1)
    Fellow eye | -2.3 (1.1) | -2.3 (1.1) | -2.3 (1.1)
Papilledema grade (fundus photography) Study Eye [Number; unit: participants] — Frisén papilledema grade is an ordinal scale that uses ocular fundus features to rate the severity of papilledema; grade 0 indicates no features of papilledema and grade 5 indicates severe papilledema.
  participants
    Study eye 1 | 8 | 12 | 20
    Study eye 2 | 32 | 23 | 55
    Study eye 3 | 20 | 20 | 40
    Study eye 4 | 24 | 21 | 45
    Study eye 5 | 2 | 3 | 5
Papilledema grade (fundus photography) Fellow eye [Number; unit: participants] — Frisén papilledema grade is an ordinal scale that uses ocular fundus features to rate the severity of papilledema; grade 0 indicates no features of papilledema and grade 5 indicates severe papilledema.
  participants
    Fellow eye 1 | 15 | 14 | 29
    Fellow eye 2 | 33 | 28 | 61
    Fellow eye 3 | 19 | 21 | 40
    Fellow eye 4 | 19 | 14 | 33
    Fellow eye 5 | 0 | 2 | 2
HIT-6 total score [Mean (Standard Deviation); unit: units on a scale] — 6-Item Headache Impact Test.
  HIT-6 total score: 36-78 (higher scores indicate greater headache severity)
  units on a scale | 60.3 (8.7) | 59.1 (9.3) | 59.7 (9.0)
CSF pressure [Mean (Standard Deviation); unit: mm H2O] — cerebrospinal fluid
  mm H2O | 348.9 (94.1) | 342.0 (70.7) | 343.5 (86.9)
SF-36 component summary score [Mean (Standard Deviation); unit: units on a scale] — Generic health-related quality of life was assessed with the 36-Item Short Form Health Survey - SF-36 consists of eight scaled scores (vitality, physical functioning bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health) : with weighted sums 0-100 (higher scores indicate better quality of life)
  units on a scale
    Physical | 45.4 (9.8) | 46.3 (8.2) | 45.8 (9.0)
    Mental | 45.2 (9.8) | 46.3 (8.2) | 45.8 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Perimetric Mean Deviation
Description: Treatment Effects on the Primary Outcome Variable, Mean change From Baseline to Month 6 in Perimetric Mean Deviation (PMD) in the Study Eye. Perimetric mean deviation is a measure of global visual field loss (mean deviation from age-corrected normal values), with a range of 2 to -32 dB; larger negative values indicate greater vision loss.
Time Frame: base line and 6 months
Population: Sixty-nine of the 86 participants (80%) in the acetazolamide group completed follow-up compared with 57 of the 79 participants (72%) in the placebo group.
Measure: Mean (Standard Error); unit: dB
Arm/Group | Acetazolamide | Sugar Pill
Number analyzed (Participants) | 69 | 57
dB | 1.43 (0.24) | 0.71 (0.28)
Statistical Analysis 1: Comparison: Acetazolamide vs Sugar Pill; Test type: Superiority or Other; p = 0.05, ANCOVA; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [0 to 1.43]

2. Secondary Outcome: Mean Change of Papilledema Grade on Fundus Photography
Description: Mean change at month 6 as compared to baseline. Frisén papilledema grade is an ordinal scale that uses ocular fundus features to rate the severity of papilledema; grade 0 indicates no features of papilledema and grade 5 indicates severe papilledema.
Time Frame: Baseline and 6 Months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acetazolamide | Sugar Pill
Number analyzed (Participants) | 69 | 57
units on a scale
  Study eye | -1.31 (0.11) | -0.61 (0.11)
  Fellow eye | -1.14 (0.10) | -0.52 (0.11)

3. Secondary Outcome: Visual Function Questionnaire (VFQ-25)
Description: Visual Function Questionnaire (VFQ-25) total score, VFQ-25 10-item neuro-ophthalmic supplement total score: 0-100 (higher scores indicate better quality of life)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetazolamide | Sugar Pill
Number analyzed (Participants) | 86 | 79
units on a scale
  Total score | 83.8 (14.1) | 82.1 (13.4)
  10-item neuro-ophthalmic supplement | 75.8 (15.4) | 75.0 (13.7)

4. Secondary Outcome: Visual Acuity (No. of Correct Letters)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: correct letters
Arm/Group | Acetazolamide | Sugar Pill
Number analyzed (Participants) | 86 | 79
correct letters
  Study Eye | 56.8 (5.1) | 55.6 (5.9)
  Fellow Eye | 58.3 (4.3) | 56.2 (6.4)

ADVERSE EVENTS:
Arm/Group | Acetazolamide | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 9/86 | 7/79
Other Adverse Events (participants affected / at risk) | 80/86 | 67/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=86) | Sugar Pill (N=79)
Rapidly failing vision (Eye disorders) | 0 | 2 (2) — Rapidly failing vision requiring hospitalization and treatment with optic nerve sheath fenestration
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0
Transaminitis (Investigations) | 1 (1) | 0
Elevated lipase with pancreatititis (Investigations) | 1 (1) | 0
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0
Allergic reaction of unknown origin (Immune system disorders) | 1 (1) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0
Pyelonephritis (Infections and infestations) | 1 (1) | 0
Live Birth (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0
Caesarean section (Surgical and medical procedures) | 1 (1) | 0
Diplopia (Ear and labyrinth disorders) | 0 | 1 (1)
Bronchitis (Infections and infestations) | 0 | 1 (1)
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 | 1 (1)
Pulmnary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 0 | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=86) | Sugar Pill (N=79)
Elevated ALT (Hepatobiliary disorders) | 6 (6) | 3 (4)
Decreased CO2 (General disorders) | 9 (9) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (14) | 3 (4)
Dizziness (General disorders) | 8 (11) | 3 (4)
Dysgeusia (General disorders) | 13 (13) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Fatigue (General disorders) | 14 (16) | 1 (1)
Headache (General disorders) | 13 (17) | 11 (16)
Nasopharyngitis (General disorders) | 5 (6) | 8 (11)
Nausea (General disorders) | 26 (30) | 10 (10)
Paresthesia (Nervous system disorders) | 41 (51) | 5 (6)
Post-LP syndrome (Surgical and medical procedures) | 5 (9) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 6 (7)
Tinnitus (Ear and labyrinth disorders) | 11 (12) | 3 (3)
Vomiting (General disorders) | 12 (13) | 3 (3)

LIMITATIONS AND CAVEATS:
A limitation is the 19% withdrawal rate which may be due, in part, to the intensity of the visit schedule. Another limitation is the difficulty in the interpretation of the estimated treatment effect on PMD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No